CLINICAL TRIAL: NCT00260585
Title: Esophageal Cancer Risk Registry
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Luketich, MD, University of Pittsburgh
Other Study IDs: STUDY19080072; NCT00260585 (Other: UPittsburgh)
Record Dates: First submitted 2005-11-28; First posted 2005-12-01 (Estimated); Last update posted 2025-04-16 (Actual); Status verified 2025-02

CONDITIONS: Esophageal Cancer; Gastroesophageal Reflux Disease (GERD); Esophageal Diseases; Hiatal Hernia; Esophageal Achalasia
Keywords: gastroesophageal reflux disease; GERD; hiatal hernia; achalasia; Barrett's metaplasia; Anti-Reflux Surgery; Known/suspected esophageal/gastroesophageal junction tumor; Esophageal disorders such as Barrett's metaplasia; Symptomatic gastroesophageal reflux disease
MeSH Terms: conditions — Esophageal Neoplasms; Gastroesophageal Reflux; Esophageal Diseases; Hernia, Hiatal; Esophageal Achalasia | interventions — Blood Specimen Collection; Tumor Burden; Biopsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, tissue, lymph nodes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Survey of client health, personal habits, family history — A questionnaire is administered at the time of consent.
Procedure: Blood specimen for non-DNA and DNA parts — Blood specimen is collected prior to surgery or at the time of scheduled routine surgical procedure(s), and at the time of routine follow-up visits
Procedure: Biopsy of esophageal/stomach tissue, lymph nodes, tumor — Tissue from the biopsies is collected intraoperatively.
Procedure: Biopsies, oral (saliva) and/or secretions, washings or mucosal scrapings/brushing from routine clinical surveillance endoscopies — Tissue from the biopsies, oral (saliva) and/or secretions, washings or mucosal scrapings/brushings are collected intraoperatively.

SUMMARY:
The purpose of this study is to identify markers in the blood and tissue that could indicate risk factors for the development and progression of esophagus cancer. This research aims to collect medical history, blood, and tissue samples from patients who present with an esophageal disorder. Identifying genetic and behavioral risk factors involved in the development of esophageal cancer might allow for early detection and prevention. Survival and an opportunity for a cure with esophageal cancer will depend greatly on the stage of diagnosis. Tumors can develop changes in their genetic (hereditary) make-up, and these changes can sometimes be seen in normal tissues before the development of cancer. These genetic (hereditary) changes can serve as tumor markers and can be detected using methods that study changes in genetic material like DNA and RNA. The analysis of proteins can provide additional information. By identifying changes in these molecules that are different or altered in cancer, the investigators can use methods and tests for the detection of these changes.

DETAILED DESCRIPTION:
We will enroll patients with esophageal cancer, patients who are at risk for developing esophageal cancer, and patients who have a non-cancerous esophageal disorder. All patients will be asked to fill out a questionnaire about their general health and personal habits, and about their relatives' medical history; this will be done during the preoperative clinic visit. Prior to or at the time of the surgical procedure(s), and at the time of routine follow-up visits, a sample of blood (about 3 tablespoons) will be drawn for research.

For patients undergoing an endoscopy after the normal biopsies are taken, several small samples will be taken from the esophagus, gastroesophageal junction, and stomach. We will also collect oral (saliva) and/or secretions, washings or mucosal scrapings/brushing from the region of the mouth, esophagus, stomach, and small bowel. In some subjects (e.g. Roux-en-y esophagojejunostomy procedure or colon interposition), secretions, washings or scrapings/brushings from the esophagus, remnant stomach, small and large bowel can also be collected. These should total no more than eight samples.

For patients undergoing an anti-reflux procedure with or without a Collis gastroplasty a lymph node is normally removed. We will receive a small piece of that lymph node after the pathologist has done the routine pathological evaluation of that node.

If the collis procedure is done, a new esophagus is formed and a small piece of stomach tissue is discarded. We will study the ordinarily discarded tissue for the transformation of cells from a normal to an abnormal state. The lymph node and stomach tissue will be collected only once for the study.

For patients undergoing an esophagectomy (removal of the esophagus) or a staging procedure (performed to determine size, exact location, and spread of tumor to nearby areas) prior to an esophagectomy small pieces of tissue will be collected (from tumor, adjacent normal esophageal lining, parts of lymph nodes, and any other tissues removed as a part of the normal procedure) from your esophagectomy or staging specimens. The samples collected will be analyzed for genetic changes in the DNA and the RNA. The samples will be stored in a locked laboratory at the Hillman Cancer Center Research Pavilion indefinitely or until the samples are depleted.

You may be contacted in the future to learn the results of any cancer screening tests you had undergone and whether anyone else in your family had developed cancer. This information will be entered in a computer data base for future study.

We may continue to collect additional blood samples and endoscopic biopsies, secretions, and scrapings during your routine clinical surveillance endoscopies. Again biopsies for normal patient management will be obtained first.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected esophageal or gastroesophageal junction malignancy
* Known Barrett's metaplasia
* Clinical management of symptomatic gastroesophageal reflux disease (GERD)
* Achalasia
* Hiatal hernia

Exclusion Criteria:

* Elevated pre-operative bloodwork will not have the additional biopsies taken.
* Platelet count less than 150,000, partial thromboplastin time (PTT) of 50 or above, and/or International Normalized Ratio (INR) of 1.8 or above will not have the additional biopsies taken.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be selected from the investigator's clinic.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 1999-06 (Actual); Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: James D. Luketich, MD, Principal Investigator — Department of Cardiothoracic Surgery
Locations (1):
- Department of Cardiothoracic Surgery, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided